CLINICAL TRIAL: NCT07249060
Title: Interferon Signature in Cancer Patients Treated With Anti-CTLA-4 and Anti-PD-1/PD-L1 Therapies: A Multicenter, Prospective, Observational Cohort Study Comparing Cancer Patients and Non-Cancer Patients With Systemic Autoimmune Diseases
Brief Title: Interferon Signature in Anti-CTLA-4 and Anti-PD-1/PD-L1-Treated Cancer Patients Compared With Systemic Autoimmune Disease Patients
Acronym: INTER-AUTENTIC
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario Araba (Other)
Collaborators: Hospital of Navarra (Other); Hospital Galdakao-Usansolo (Other Government); Hospital San Pedro de Logroño (Other); Consorci Sanitari del Maresme. Hospital Universitari de Mataró (Other); Hospital Donostia (Other)
Responsible Party: Principal Investigator, Iñigo Les Bujanda, Iñigo Les Bujanda, Hospital of Navarra
Other Study IDs: PI_2023/90
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Immune-Related Adverse Events; Lupus Erythematosus, Systemic; Sjogren Syndrome; Systemic Sclerosis (SSc); Inflammatory Myopathies; Solid Tumors
Keywords: Immune Checkpoint Inhibitors; Adverse events; Biomarkers; Predictive; Prospective Studies; Immune System
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Scleroderma, Systemic; Myositis | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Biospecimen Retention: Samples With DNA — The specific types of biospecimens that will be retained are serum and buffy coat.
  * Serum: Six aliquots of 500 μL will be processed and stored from each sample at every collection time point.
  * Buffy Coat: Two tubes of buffy coat will be retained from each sample (one tube will contain RNAlater for subsequent RNA isolation); however, this specific biospecimen will only be processed and collected during the V1, V5, and V7 treatment cycles.
  All collected samples will be kept frozen at -80°C and stored in a coded manner to maintain confidentiality and sample integrity for future approved research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICI cohort: Patients with cancer treated with immune checkpoint inhibitors
  Interventions: Drug: Immune Checkpoint Inhibitors
- SAD cohort: Patients without cancer affected by systemic lupus erythematosus, primary Sjögren's syndrome, progressive systemic sclerosis, and/or idiopathic inflammatory myopathy.

INTERVENTIONS:
Drug: Immune Checkpoint Inhibitors — Administration of immune checkpoint inhibitors according to protocol
  Groups: ICI cohort

SUMMARY:
This study aims to identify a way to predict the side effects that some people with cancer experience when receiving immunotherapy. These side effects, known as immune-related adverse events (irAEs), occur when the immune system mistakenly attacks healthy tissues, like certain autoimmune diseases. At present, clinicians lack reliable tests to determine who is most likely to develop these reactions. The goal of this study is to determine whether substances in the blood called interferons (IFNs) could serve as early warning markers.

The study will include 300 people with cancer who are about to begin immunotherapy. To provide a meaningful comparison, the investigators will also enroll 40 individuals with autoimmune diseases such as lupus. Understanding how IFN levels differ between these groups may help clarify whether IFN patterns in cancer patients resemble those seen in autoimmune disease.

Participants in both groups will be asked to provide small blood samples at predefined time points during their clinical care or treatment. Researchers will measure the levels of different IFN types in all samples to compare IFN levels between cancer patients and individuals with autoimmune diseases, and within the cancer group between patients who develop irAEs and those who do not. The long-term aim of the study is to develop a simple test that can help clinicians identify patients at higher risk of irAEs.

Immune-related adverse events (irAEs) are a frequent complication in cancer patients treated with immune checkpoint inhibitors (ICIs), and they often resemble or exacerbate preexisting autoimmune diseases. Despite extensive research in the field, no validated predictive biomarkers of irAEs currently exist. Emerging evidence suggests that the IFN signature -long implicated in the pathogenesis of several systemic autoimmune diseases (SADs)- may also be upregulated in patients who develop ICI-induced irAEs, likely with substantial overlap among different IFN subtypes. Given these clinical and molecular similarities with SADs, it is plausible that IFN levels in peripheral blood carry predictive value for irAE risk, although the dominant IFN types in ICI-related toxicity remain unknown.

The INTER-AUTENTIC project aims to determine whether baseline IFN levels and their dynamic changes, measured in peripheral blood using a dedicated panel, can predict the onset of irAEs in cancer patients receiving ICIs. Supported by the Medical Oncology departments of six university hospitals in Northern Spain, this multicenter, observational, prospective cohort study has been underway since 2021. Biobank samples have been collected from ICI-treated patients before treatment initiation, at protocol-defined time points, and at the moment of irAE diagnosis (ICI cohort). The study seeks to identify the IFN subtypes with the most pronounced differential expression between patients with and without irAEs, and to evaluate whether IFN levels enhance the predictive performance of a model incorporating other clinical variables potentially associated with immune-mediated toxicity. A sample size of 300 cancer patients has been estimated for this analysis.

In addition, a second prospective cohort of 40 non-cancer patients with systemic lupus erythematosus, primary Sjögren's syndrome, systemic sclerosis, and/or idiopathic inflammatory myopathy (SAD cohort) will be included. Since IFNs play a well-established pathogenic role in these conditions, this cohort will allow characterization of the IFN signature at key follow-up points (baseline, remission, and disease flare) and comparison with the IFN profiles of ICI-treated patients, regardless of whether they develop irAEs.

ELIGIBILITY:
ICI cohort:

Inclusion Criteria:

* Initiation of treatment with a single ICI or dual ICI therapy in accordance with current clinical guidelines;
* Patients who are treatment-naïve to ICIs; and
* Age ≥18 years.

Exclusion Criteria:

* Estimated mortality of less than 3 months from the start of treatment;
* Current combination therapy with chemotherapy, tyrosine kinase inhibitors, or other tumor-specific treatments;
* Contraindication to treatment with ICIs (documented hypersensitivity, severe active autoimmune disease, Eastern Cooperative Oncology Group [ECOG] ≥3);
* Ongoing immunosuppressive therapy, including prednisone at doses >10 mg/day or equivalent.

SAD cohort:

Inclusion Criteria:

* Meeting classification criteria for Systemic Lupus Erythematosus (SLE) (ACR/EULAR 2019), Primary Sjögren's Syndrome (pSS) (ACR/EULAR 2016), Systemic Sclerosis (SSc) (ACR/EULAR 2013), and/or Idiopathic Inflammatory Myopathy (IIM) (ACR/EULAR 2017).
* Age ≥18 years old.

Exclusion Criteria:

* Estimated mortality less than 3 months from the start of follow-up.
* Active immunosuppressive treatment, including prednisone at doses >10 mg/day or equivalent.
* Recent diagnosis (<1 year) of cancer, with the exception of non-melanoma skin cancer, or currently receiving active oncology-specific treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICI cohort: Patients in the ICI cohort will be recruited from the Medical Oncology outpatient clinics of the participating hospitals. All patients diagnosed with a solid neoplasm eligible for treatment with ICIs will be considered for inclusion, using consecutive case sampling.
  SAD cohort: Patients in the SAD cohort will be recruited in the outpatient clinics of the HUN Internal Medicine Service's SAD Unit, using consecutive case sampling.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of immune-related adverse event | 48 weeks
  any symptom, sign, syndrome, or disease caused by an immune-activating mechanism during the administration of an ICI once other causes such as an infectious disease or tumor progression have been ruled out.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Les I, Perez-Francisco I, Cabero M, Sanchez C, Hidalgo M, Teijeira L, Arrazubi V, Dominguez S, Anaut P, Eguiluz S, Elejalde I, Herrera A, Martinez M. Prediction of Immune-Related Adverse Events Induced by Immune Checkpoint Inhibitors With a Panel of Autoantibodies: Protocol of a Multicenter, Prospective, Observational Cohort Study. Front Pharmacol. 2022 Jun 1;13:894550. doi: 10.3389/fphar.2022.894550. eCollection 2022. PMID 35721217
- [Background] Riudavets M, Mosquera J, Garcia-Campelo R, Serra J, Anguera G, Gallardo P, Sullivan I, Barba A, Del Carpio L, Barnadas A, Gich I, Majem M. Immune-Related Adverse Events and Corticosteroid Use for Cancer-Related Symptoms Are Associated With Efficacy in Patients With Non-small Cell Lung Cancer Receiving Anti-PD-(L)1 Blockade Agents. Front Oncol. 2020 Sep 7;10:1677. doi: 10.3389/fonc.2020.01677. eCollection 2020. PMID 33014837
- [Background] Hailemichael Y, Johnson DH, Abdel-Wahab N, Foo WC, Bentebibel SE, Daher M, Haymaker C, Wani K, Saberian C, Ogata D, Kim ST, Nurieva R, Lazar AJ, Abu-Sbeih H, Fa'ak F, Mathew A, Wang Y, Falohun A, Trinh V, Zobniw C, Spillson C, Burks JK, Awiwi M, Elsayes K, Soto LS, Melendez BD, Davies MA, Wargo J, Curry J, Yee C, Lizee G, Singh S, Sharma P, Allison JP, Hwu P, Ekmekcioglu S, Diab A. Interleukin-6 blockade abrogates immunotherapy toxicity and promotes tumor immunity. Cancer Cell. 2022 May 9;40(5):509-523.e6. doi: 10.1016/j.ccell.2022.04.004. Epub 2022 May 9. PMID 35537412
- [Background] Bishu S, Melia J, Sharfman W, Lao CD, Fecher LA, Higgins PDR. Efficacy and Outcome of Tofacitinib in Immune checkpoint Inhibitor Colitis. Gastroenterology. 2021 Feb;160(3):932-934.e3. doi: 10.1053/j.gastro.2020.10.029. Epub 2020 Oct 21. No abstract available. PMID 33096100
- [Background] Fernandez-Ruiz R, Niewold TB. Type I Interferons in Autoimmunity. J Invest Dermatol. 2022 Mar;142(3 Pt B):793-803. doi: 10.1016/j.jid.2021.11.031. Epub 2022 Jan 10. PMID 35016780
- [Background] Unger JM, Vaidya R, Albain KS, LeBlanc M, Minasian LM, Gotay CC, Henry NL, Fisch MJ, Lee SM, Blanke CD, Hershman DL. Sex Differences in Risk of Severe Adverse Events in Patients Receiving Immunotherapy, Targeted Therapy, or Chemotherapy in Cancer Clinical Trials. J Clin Oncol. 2022 May 1;40(13):1474-1486. doi: 10.1200/JCO.21.02377. Epub 2022 Feb 4. PMID 35119908
- [Background] Wang M, Zhai X, Li J, Guan J, Xu S, Li Y, Zhu H. The Role of Cytokines in Predicting the Response and Adverse Events Related to Immune Checkpoint Inhibitors. Front Immunol. 2021 Jul 22;12:670391. doi: 10.3389/fimmu.2021.670391. eCollection 2021. PMID 34367136
- [Background] Traves PG, Murray B, Campigotto F, Galien R, Meng A, Di Paolo JA. JAK selectivity and the implications for clinical inhibition of pharmacodynamic cytokine signalling by filgotinib, upadacitinib, tofacitinib and baricitinib. Ann Rheum Dis. 2021 Jul;80(7):865-875. doi: 10.1136/annrheumdis-2020-219012. Epub 2021 Mar 19. PMID 33741556
- [Background] Coukos A, Vionnet J, Obeid M, Bouchaab H, Peters S, Latifyan S, Wicky A, Michielin O, Chtioui H, Moradpour D, Fasquelle F, Sempoux C, Fraga M. Systematic comparison with autoimmune liver disease identifies specific histological features of immune checkpoint inhibitor-related adverse events. J Immunother Cancer. 2022 Oct;10(10):e005635. doi: 10.1136/jitc-2022-005635. PMID 36283734
- [Background] Pinal-Fernandez I, Quintana A, Milisenda JC, Casal-Dominguez M, Munoz-Braceras S, Derfoul A, Torres-Ruiz J, Pak K, Dell'Orso S, Naz F, Gutierrez-Cruz G, Milone M, Shelly S, Duque-Jaimez Y, Tobias-Baraja E, Matas-Garcia A, Garrabou G, Padrosa J, Ros J, Trallero-Araguas E, Walitt B, Christopher-Stine L, Lloyd TE, Zhao C, Swift S, Rajan A, Grau-Junyent JM, Selva-O'Callaghan A, Liewluck T, Mammen AL. Transcriptomic profiling reveals distinct subsets of immune checkpoint inhibitor induced myositis. Ann Rheum Dis. 2023 Jun;82(6):829-836. doi: 10.1136/ard-2022-223792. Epub 2023 Feb 17. PMID 36801811
- [Background] Salem JE, Bretagne M, Abbar B, Leonard-Louis S, Ederhy S, Redheuil A, Boussouar S, Nguyen LS, Procureur A, Stein F, Fenioux C, Devos P, Gougis P, Dres M, Demoule A, Psimaras D, Lenglet T, Maisonobe T, De Chambrun MP, Hekimian G, Straus C, Gonzalez-Bermejo J, Klatzmann D, Rigolet A, Guillaume-Jugnot P, Champtiaux N, Benveniste O, Weiss N, Saheb S, Rouvier P, Plu I, Gandjbakhch E, Kerneis M, Hammoudi N, Zahr N, Llontop C, Morelot-Panzini C, Lehmann L, Qin J, Moslehi JJ, Rosenzwajg M, Similowski T, Allenbach Y. Abatacept/Ruxolitinib and Screening for Concomitant Respiratory Muscle Failure to Mitigate Fatality of Immune-Checkpoint Inhibitor Myocarditis. Cancer Discov. 2023 May 4;13(5):1100-1115. doi: 10.1158/2159-8290.CD-22-1180. PMID 36815259
- [Background] Soret P, Le Dantec C, Desvaux E, Foulquier N, Chassagnol B, Hubert S, Jamin C, Barturen G, Desachy G, Devauchelle-Pensec V, Boudjeniba C, Cornec D, Saraux A, Jousse-Joulin S, Barbarroja N, Rodriguez-Pinto I, De Langhe E, Beretta L, Chizzolini C, Kovacs L, Witte T; PRECISESADS Clinical Consortium; PRECISESADS Flow Cytometry Consortium; Bettacchioli E, Buttgereit A, Makowska Z, Lesche R, Borghi MO, Martin J, Courtade-Gaiani S, Xuereb L, Guedj M, Moingeon P, Alarcon-Riquelme ME, Laigle L, Pers JO. A new molecular classification to drive precision treatment strategies in primary Sjogren's syndrome. Nat Commun. 2021 Jun 10;12(1):3523. doi: 10.1038/s41467-021-23472-7. PMID 34112769
- [Background] Henderson Berg MH, Del Rincon SV, Miller WH. Potential therapies for immune-related adverse events associated with immune checkpoint inhibition: from monoclonal antibodies to kinase inhibition. J Immunother Cancer. 2022 Jan;10(1):e003551. doi: 10.1136/jitc-2021-003551. PMID 35086945
- [Background] Nunez NG, Berner F, Friebel E, Unger S, Wyss N, Gomez JM, Purde MT, Niederer R, Porsch M, Lichtensteiger C, Kramer R, Erdmann M, Schmitt C, Heinzerling L, Abdou MT, Karbach J, Schadendorf D, Zimmer L, Ugurel S, Klumper N, Holzel M, Power L, Kreutmair S, Capone M, Madonna G, Cevhertas L, Heider A, Amaral T, Hasan Ali O, Bomze D, Dimitriou F, Diem S, Ascierto PA, Dummer R, Jager E, Driessen C, Levesque MP, van de Veen W, Joerger M, Fruh M, Becher B, Flatz L. Immune signatures predict development of autoimmune toxicity in patients with cancer treated with immune checkpoint inhibitors. Med. 2023 Feb 10;4(2):113-129.e7. doi: 10.1016/j.medj.2022.12.007. Epub 2023 Jan 23. PMID 36693381
- [Background] Les I, Martinez M, Perez-Francisco I, Cabero M, Teijeira L, Arrazubi V, Torrego N, Campillo-Calatayud A, Elejalde I, Kochan G, Escors D. Predictive Biomarkers for Checkpoint Inhibitor Immune-Related Adverse Events. Cancers (Basel). 2023 Mar 6;15(5):1629. doi: 10.3390/cancers15051629. PMID 36900420
- [Background] Ramos-Casals M, Brahmer JR, Callahan MK, Flores-Chavez A, Keegan N, Khamashta MA, Lambotte O, Mariette X, Prat A, Suarez-Almazor ME. Immune-related adverse events of checkpoint inhibitors. Nat Rev Dis Primers. 2020 May 7;6(1):38. doi: 10.1038/s41572-020-0160-6. PMID 32382051
- [Background] Haslam A, Gill J, Prasad V. Estimation of the Percentage of US Patients With Cancer Who Are Eligible for Immune Checkpoint Inhibitor Drugs. JAMA Netw Open. 2020 Mar 2;3(3):e200423. doi: 10.1001/jamanetworkopen.2020.0423. PMID 32150268